CLINICAL TRIAL: NCT06087159
Title: Promoting Mental Health of Teachers and Caregivers Using a Personalized mHealth Toolkit in Uganda
Brief Title: Promoting Mental Health of Teachers and Caregiver Using a Personalized mHealth Toolkit in Uganda
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-00600
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Mental Health Literacy; Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mWEL Intervention (Phase 1 and Phase 2) (Experimental): Teachers or parents of children in participating schools who are randomly assigned to receive the mWEL intervention.
  Interventions: Behavioral: mHealth Toolkit for Wellness & Empowering Lives of School Community (mWEL)
- Control (Phase 1 and Phase 2) (No Intervention): Teachers or parents of children in participating schools who are randomly assigned to the control arm.

INTERVENTIONS:
Behavioral: mHealth Toolkit for Wellness & Empowering Lives of School Community (mWEL) — mWEL-App is a preventive intervention tool for teachers and parents as a self-help support. It integrates three key mental health presentive service functions: i) comprehensive screen to assess mental health (anxiety, depression), stress, and related contextual risks; ii) a tailored strength and weakness profile/report with recommendations to promote self-awareness and mental health knowledge; and iii) tailored evidence-based strategies and additional support and clinical resources to improve skills in stress management, emotion regulation, and maintain mental wellness. mWEL will be designed as a self-administered tool. Participating parents and teachers can access to mWEL app after they sign up for an account. Intervention participants will have access to the App anytime within a 3-5 month study period.
  Arms: mWEL Intervention (Phase 1 and Phase 2)

SUMMARY:
This study record describes a two-phase of clinical trial study. The first phase is a pilot study phase (to study feasibility and efficacy of the intervention), and the second phase is an effectiveness study phase (a fully powered evaluation study to test the intervention effectiveness). This proposal seeks to develop and test a new mHealth intervention, the mHealth Toolkit for Wellness & Empowering Lives of School Community (mWEL) in Uganda. The mWEL-digial toolkit is a preventive intervention tool for teachers and parents as a self-help support modality. Caregivers who need support in navigating the toolkit will be supported by peer-community health workers (P-CHWs).

DETAILED DESCRIPTION:
During the first phase (from 11-01-2024 to 8-15-2025), a cluster randomized controlled trial (cRCT) with 8 schools (4 intervention and 4 wait-list control schools) including 160 caregivers (80 teachers and 80 parents) is conducted. The aim of the pilot RCT is to pilot test the implementation process, feasibility, acceptability, usage patterns, and efficacy of the mWEL. The investigators hypothesize that: 1) relative to the control, caregivers receiving the mWEL will have better efficacy outcomes (mental health literacy, and mental health outcomes); and 2) mWEL implementation will have high acceptability, appropriateness, and feasibility.

During the second phase (from 10-01-2025 to 08-31-2028), the optimized version of mWEL toolkit will be further tested for effectiveness using a cRCT and a matched-pair randomization method. The sample will be recruited from urban and rural schools. In intervention schools, participants will engage with the mWEL toolkit through group sessions or one-on-one support with Peer-Community Health Workers (P-CHWs). Control schools will receive general and non-mental health related health literacy information, and without any tailored support. Impacts on caregivers' health literacy and their mental health (anxiety, depression) will be evaluated (n=1000, 500 parents and 500 teachers in 24 schools, with 12 intervention and 12 wait-list control). The investigators hypothesize that: 1) relative to control, teachers and parents receiving mWEL will have better effectiveness outcomes (i.e., mental health literacy, and mental health outcomes; and 2) similar effectiveness findings for urban/rural schools and for male/female.

ELIGIBILITY:
Teachers Inclusion Criteria:

* Teaching in recruited schools.
* At least 18 years old.

Parents Inclusion Criteria:

* At least 18 years old.
* Have a child aged 6-14 years.

Exclusion Criteria:

* Evidence of psychopathology or cognitive impairment severe enough to preclude giving consent, or completing the survey instruments or the focus group of the study.
* Parents/Teachers/Caregivers who are not in one of our recruited primary school
* Participants under the age of 18
* Participant who does not speak English and Luganda will not be able to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1180 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Universal Mental Health Literacy Scale Score | Baseline, Month 5
  The Universal Mental Health Literacy Scale comprises 21 items asking respondents to indicate their knowledge of various aspects regarding mental health. Items are rated on Yes/No or 5-point Likert scales. The total score is produced by mean of all item scores and ranges from 1-5 or % correct knowledge; higher scores indicate greater mental health literacy
Change in PHQ-9 Score | Baseline, Month 5
  The Patient Health Questionnaire-9 (PHQ-9) is a widely used self-administered tool designed to screen, diagnose, and monitor the severity of depression in individuals. It consists of nine questions that align directly with the diagnostic criteria for major depressive disorder in the DSM-5. Each item asks about the frequency of specific depressive symptoms experienced over the past two weeks (on a 0 to 3 point Likert scales), such as low mood, loss of interest, sleep problems, fatigue, appetite changes, feelings of worthlessness, trouble concentrating, psychomotor changes, and thoughts of self-harm or suicide. The total score ranges from 0 to 27, with higher scores indicating more severe depression. Severity is typically interpreted as follows:
  0-4: None to minimal depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20-27: Severe depression
Change in GAD-7 Anxiety Score | Baseline, Month 5
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a brief, self-administered questionnaire designed to screen for and assess the severity of generalized anxiety disorder (GAD) symptoms over the past two weeks. The scale is rated on a 0 to 3 point Likert scales). The total GAD-7 score ranges from 0 to 21, with higher scores indicating greater anxiety severity. Severity is commonly interpreted as:
  0-4: Minimal anxiety 5-9: Mild anxiety 10-14: Moderate anxiety 15-21: Severe anxiety
  Less than 55 = None to slight depression 55.0-59.9 = Mild depression 60.0-69.9 = Moderate depression 70 and over = Severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Keng-Yen Huang, PhD, MPH, Principal Investigator — NYU Langone Health
Locations (2):
- Uganda (2):
  - Study Site, Kampala
  - Study Site, Nakaseke

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Keng-Yen.Huang@nyulangone.org The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Keng-Yen.Huang@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2024-12-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT06087159/ICF_000.pdf